CLINICAL TRIAL: NCT06055686
Title: The Use of Electrical Stimulation for Determination of Epidural Catheter Placement
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor-Med Ctr Line, Stanford University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 71662
Record Dates: First submitted 2023-09-20; First posted 2023-09-28 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Obstetric Pain; Anesthesia, Local
Keywords: Electrical Epidural Stimulation Test; Epidural Failure
MeSH Terms: conditions — Labor Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Electrical Epidural Stimulation Test (Experimental): Laboring women who request epidural analgesia will be given an electric stimulation at incremental points during catheter pull back with documentation of where stimulation was seen.
  Interventions: Diagnostic Test: Electrical Epidural Stimulation Test

INTERVENTIONS:
Diagnostic Test: Electrical Epidural Stimulation Test — Electrical stimulation test measures sensory/motor responses

SUMMARY:
The aim of this study is to address the problem of epidural failure. The investigators theorize epidural failure can be due to inappropriate catheter movement and this may be related to the length of which the epidural catheter is inserted. The investigators will use electrical stimulation to determine if the catheter moved in the sacral direction with insertion.

DETAILED DESCRIPTION:
The research participants will be pregnant women in Labor and Delivery ward of Stanford University hospital who request an epidural for labor analgesia.

In this study the patients will receive an epidural catheter in the same way as standard of care. The catheter will be inserted to 20cm and then electrically stimulated to document where it is placed by looking at the muscles effected. The catheter is then pulled back in 5cm increments and stimulated until the standard distance is achieved. For example, if loss of resistance happened at 5cm, the catheter would be inserted to 20cm, stimulated, pulled back to 15cm and stimulated, and finally to 10cm and stimulated.

Electrical stimulation of epidural catheters for confirmation of placement is a published and accepted technique. In this study, the investigators will perform electrical stimulation at incremental points during catheter pull back with documentation of where stimulation was seen.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant female requesting epidural for labor analgesia.
* Must meet standard inclusion criteria for safe epidural placement.
* Platelet count over 70,000, INR under 1.3.

Exclusion Criteria:

* Unable to safely place epidural catheter due to commonly accepted patient factors.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2026-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Incidence rate of sacral stimulation | 1 year
  Electrical stimulation will be performed at incremental points during catheter pull back with documentation of where stimulation was seen.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Abboud, MD, Study Director — Clinical Instructor, Anesthesiology, Perioperative and Pain Medicine
Locations (1):
- Lucile Packard Childrens Hospital, Stanford, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim YS, Kim HS, Jeong H, Lee CH, Lee MK, Choi SS. Efficacy of electrical stimulation on epidural anesthesia for cesarean section: a randomized controlled trial. BMC Anesthesiol. 2020 Jun 10;20(1):146. doi: 10.1186/s12871-020-01063-1. PMID 32522156
- [Background] Charghi R, Chan SY, Kardash KJ, Finlayson RJ, Tran DQ. Electrical stimulation of the epidural space using a catheter with a removable stylet. Reg Anesth Pain Med. 2007 Mar-Apr;32(2):152-6. doi: 10.1016/j.rapm.2006.10.006. PMID 17350527
- [Background] Kwofie MK, Launcelott G, Tsui BCH. Determination of thoracic epidural catheter placement: electrical epidural stimulation (Tsui test) is simple, effective, and under-utilized. Can J Anaesth. 2019 Apr;66(4):360-364. doi: 10.1007/s12630-019-01302-1. Epub 2019 Jan 23. No abstract available. PMID 30675686